CLINICAL TRIAL: NCT01958645
Title: A Phase I, Single-blind, Randomised, Placebo-controlled, Single Centre Study to Investigate the Safety, Tolerability and Pharmacodynamics of Intravenous MEDI8111 After Single Ascending Doses in Healthy Male Subjects
Brief Title: To Assess Safety, Tolerability and Pharmacodynamics of Intravenous MEDI8111 After Single Ascending Doses.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D5050C00001
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Subjects
Keywords: Phase 1, healthy male subjects, safety and tolerability, pharmacodynamic, pharmacokinetic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): MEDI8111
  Interventions: Drug: MEDI8111
- B (Placebo Comparator): Placebo for MEDI8111
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MEDI8111 — MEDI8111 lyophilisate for solution for infusion
  Arms: A
Other: Placebo — Placebo for MEDI8111 saline solution for infusion
  Arms: B

SUMMARY:
A study to investigate the safety, tolerability and pharmacodynamics of MEDI8111 after single ascending doses in healthy male.

DETAILED DESCRIPTION:
A phase I, single-blind, randomised, placebo-controlled, single centre study to investigate the safety, tolerability and pharmacodynamics of intravenous MEDI8111 after single ascending doses in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures, Healthy male subjects aged 18-40 years with suitable veins for cannulation or repeated venepuncture, Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weight at least 50 kg an no more than 100 kg inclusive, Male subjects should be willing to avoid fathering a child by either true abstinence or the use of two effective means of contraception from the day of dosing until 3 months after dosing with the IP. They should also be willing to use barrier methods from the day of dosing until 3 months after dosing.

Exclusion Criteria:

* Prothrombotic mutation such as factor V Leiden, or deficiencies of protein C, protein S, prothrombin, antithrombin or APC, Antibodies to coagulation FII, History or family history of venous or arterial thromboembolic event, and/or myocardial infarction before age of 50 years, ETP level at baseline >2000nM/min, FII level (by clot) at screening and/or at baseline outside 50-250% of the normal range

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Wahlander, MD, Study Director — AstraZeneca Mölndal, Sweden; Anders Berggren, MD, Study Chair — AstraZeneca Mölndal, Sweden; Timothy Mant, Prof, Principal Investigator — Quintiles London, United Kingdom
Locations (1):
- Research Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male healthy volunteers recruited by advertisement during the period October 2013 - October 2014
Pre-assignment Details: The study was prematurely terminated after 2 cohorts as dose escalation stopping criteria (PD thresholds) were reached and it was judged to be of limited value to expose more healthy subjects.
  Cohort 1: 2 placebo + 4 MEDI8111 dose 1. Cohort 2: 2 placebo + 4 MEDI8111 dose 2.
Groups:
- Placebo: Placebo (Saline solution for infusion)
- MEDI8111 Dose 1: MEDI8111 dose 1 (Lyophilisate for solution for infusion, 30 mg)
- MEDI8111 Dose 2: MEDI8111 dose 2 (Lyophilisate for solution for infusion, 30 mg)
Period: Overall Study
Arm/Group | Placebo | MEDI8111 Dose 1 | MEDI8111 Dose 2
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI8111 Dose 1 | MEDI8111 Dose 2 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (9) | 30 (6) | 30 (6) | 29 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 2 | 3 | 3 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Description of the Safety Profile in Terms of Adverse Events (AE),Vital Signs, ECG, Lab Variables, Immunogenicity and Physical Examination
Time Frame: From screening and up to the lab follow-up visit (Day 29)
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI8111 Dose 1 | MEDI8111 Dose 2
Number analyzed (Participants) | 4 | 4 | 4
Participants
  Subjects with any AE | 2 | 3 | 2
  Gastrointestinal disorders | 1 | 1 | 1
  Infections and infestations | 0 | 1 | 1
  Investigations | 0 | 1 | 0
  Musculoskeletal and connective tissue disorders | 0 | 1 | 0
  Nervous system disorder | 0 | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 1 | 0 | 1
  Skin and subcutaneous tissue disorders | 1 | 0 | 0

2. Secondary Outcome: Change From Baseline Endogenous Thrombin Potential (ETP)
Description: For the baseline variables and adverse events the two placebo arms (placebo dose 1 and placebo dose 2) are recorded as one. For the secondary outcome measures the two placebo arms are recorded separately.
Time Frame: Predose and Days 1-5
Measure: Mean (Standard Deviation); unit: nM*min
Groups:
- Placebo Dose 1: Placebo dose 1 (Saline solution for infusion)
- Placebo Dose 2: Placebo dose 2 (Saline solution for infusion)
Arm/Group | Placebo Dose 1 | MEDI8111 Dose 1 | MEDI8111 Dose 2 | Placebo Dose 2
Number analyzed (Participants) | 2 | 4 | 4 | 2
nM*min
  0.98 h | 16 (143) | 131 (219) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  1.03 h | 30.5 (138) | 145 (263) | 39.8 (72.1) | -35.0 (214)
  1.25 h | 67.0 (356) | 135 (345) | 211 (179) | 27.0 (80.6)
  1.5 h | 166 (75) | -17.3 (120) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  2 h | 32.5 (148) | 178 (336) | 147 (167) | -79.5 (95.5)
  3 h | 57.0 (238) | 188 (385) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  4 h | -88.0 (226) | 72.8 (545) | 157 (277) | 4.50 (48.8)
  8 h | 157 (161) | 141 (288) | 83.0 (216) | 6.50 (33.2)
  12 h | 82.5 (70.0) | 366 (396) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  24 h | -29.0 (279) | 115 (336) | 86.0 (120) | 70.5 (14.8)
  36 h | -59.0 (134) | 329 (496) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  48 h | 29.0 (222) | 172 (264) | 206 (261) | 91.0 (26.9)
  72 h | 183 (222) | 71.5 (274) | 139 (194) | 73.5 (9.19)
  96 h | -95.0 (209) | -1.00 (483) | 64.8 (223) | 46.0 (8.49)
  Follow up | -12.5 (13.4) | -34.5 (206) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.

3. Secondary Outcome: Change From Baseline Factor II Concentrations by ECL Assay
Time Frame: Predose and 1-8 hours
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo Dose 1 | MEDI8111 Dose 1 | MEDI8111 Dose 2 | Placebo Dose 2
Number analyzed (Participants) | 2 | 4 | 4 | 2
umol/L
  0.33 h | -0.0810 (0.0410) | -0.0188 (0.0661) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  0.67 h | -0.0480 (0.0113) | 0.0275 (0.0377) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  0.98 h | -0.134 (0.0368) | 0.00450 (0.0896) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  1 h | -0.131 (0.0156) | -0.0305 (0.0435) | 0.166 (0.0632) | 0.0650 (0.0212)
  1.25 h | -0.143 (0.00354) | -0.0920 (0.0881) | 0.116 (0.113) | 0.0600 (0.0424)
  1.5 h | -0.132 (0.121) | -0.124 (0.148) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  2 h | -0.0655 (0.0629) | 0.00450 (0.188) | 0.111 (0.129) | 0.0800 (0.0849)
  3 h | -0.0675 (0.248) | 0.0608 (0.120) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  4 h | -0.127 (0.279) | 0.123 (0.0663) | 0.141 (0.155) | 0.0450 (0.0495)
  8 h | 0.00650 (0.122) | 0.0633 (0.0801) | 0.0835 (0.0731) | -0.00900 (0.0410)

4. Secondary Outcome: Change From Baseline Factor II Concentrations by Clot Assay
Time Frame: Predose and 1-8 hours
Measure: Mean (Standard Deviation); unit: % (concentration)
Arm/Group | Placebo Dose 1 | MEDI8111 Dose 1 | MEDI8111 Dose 2 | Placebo Dose 2
Number analyzed (Participants) | 2 | 4 | 4 | 2
% (concentration)
  0.33 h | 7.65 (26.4) | -1.40 (7.67) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  0.67 h | 3.15 (17.2) | 1.35 (6.95) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  0.98 h | -9.35 (12.2) | -2.40 (4.25) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  1 h | -14.4 (13.6) | -1.15 (4.22) | 13.7 (14.5) | 7.30 (0.00)
  1.25 | -6.85 (18.6) | -0.400 (5.54) | 12.2 (9.55) | 8.30 (1.41)
  1.5 h | -10.9 (12.9) | -0.400 (8.67) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  2 h | -8.85 (8.70) | 0.350 (5.45) | 10.5 (7.84) | 2.80 (4.95)
  3 h | -5.85 (12.9) | 1.10 (9.73) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  4 h | 0.150 (15.8) | 2.10 (4.45) | 18.2 (9.02) | 7.30 (4.24)
  8 h | -9.85 (10.1) | -1.90 (5.78) | 11.7 (9.12) | 9.30 (4.24)

5. Secondary Outcome: Change From Baseline D-dimer Concentration
Time Frame: predose and 1-8 hours
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo Dose 1 | MEDI8111 Dose 1 | MEDI8111 Dose 2 | Placebo Dose 2
Number analyzed (Participants) | 2 | 4 | 4 | 2
mg/L
  0.98 h | -0.0169 (0.0144) | 0.0408 (0.103) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  1.03 h | 0.0432 (0.0564) | 0.0383 (0.109) | 0.0108 (0.0190) | 0.0270 (0.0141)
  1.25 h | 0.0232 (0.113) | 0.000750 (0.0336) | 0.0333 (0.0306) | 0.0170 (0.0566)
  1.5 h | -0.00185 (0.0214) | 0.408 (0.795) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  2 h | 0.0682 (0.135) | 0.0382 (0.0813) | 0.0610 (0.0760) | 0.0170 (0.0424)
  3 h | 0.0732 (0.0846) | 0.00325 (0.0237) | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point.
  4 h | NA (NA) — No sample was planned to be collected at this time point. | NA (NA) — No sample was planned to be collected at this time point. | 0.0933 (0.0810) | 0.207 (0.0849)
  8 h | 0.588 (0.799) | 0.0858 (0.0914) | 0.0633 (0.0630) | 0.0470 (0.0849)

ADVERSE EVENTS:
Time Frame: At screening, Days 1-5
Arm/Group | Placebo | MEDI8111 Dose 1 | MEDI8111 Dose 2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 3/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | MEDI8111 Dose 1 (N=4) | MEDI8111 Dose 2 (N=4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Fibrin D-dimer increased (Investigations) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Limitations: few subjects, high variability of coagulation variables

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No